CLINICAL TRIAL: NCT05456542
Title: Cuff Leak Test and Airway Obstruction in Mechanically Ventilated ICU Patients (COSMIC): A Pilot Randomized Controlled Trial
Brief Title: Cuff Leak Test and Airway Obstruction in Mechanically Ventilated ICU Patients
Acronym: COSMIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Principal Investigator, Kimberley Lewis, Principal Investigator, SJHH Staff Intensivist, Assistant Professor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 3480
Record Dates: First submitted 2022-05-03; First posted 2022-07-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Failure
Keywords: Laryngeal Edema, Mechanical Ventilation, Cuff Leak Test
MeSH Terms: conditions — Respiratory Insufficiency; Laryngeal Edema | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Multicentred, national, parallel-group, pragmatic vanguard pilot trial.
Who Masked: Outcomes Assessor
Masking Description: The Research Coordinator will randomize eligible patients in a 1:1 allocation using undisclosed variable block sizes through a central computer system on REDCap. Randomization algorithm will stratify patients by recruitment site. This is an unblinded study as group allocation will be known. However, outcome adjudicators and the study statistician will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - Cuff Leak Test (Experimental): A respiratory therapist will perform a Cuff Leak Test on all patients prior to extubation. If no air leak is auscultated (a failed CLT), extubation will be delayed. During this time, the patient will receive dexamethasone 4mg intravenous every 6 hours for 12-24 hours and the clinical team will be advised to consider optimizing a patient's fluid status through either diuresis or ultrafiltration if the patient has renal failure. After 12-24 hours, and once the clinical team decides the patient is ready for another extubation attempt, the CLT will be repeated. If the patient fails the CLT again, it will be at the discretion of the clinical team how to proceed (i.e. continue steroid administration, and further delay extubation vs immediately extubating despite a failed CLT) (Figure 3). A passed CLT at any time point will result in immediate extubation.
  Interventions: Diagnostic Test: Cuff Leak Test; Drug: Dexamethasone 4mg
- Control - No Cuff Leak Test (No Intervention): In the control group, once the patient is deemed ready for extubation by the clinical team, the patient will be extubated without performing a CLT, without administration of corticosteroids, and without delay.

INTERVENTIONS:
Diagnostic Test: Cuff Leak Test — Clinicians perform the cuff leak test (CLT) to help optimize extubation. The test requires deflation of the cuff at the end of the endotracheal tube (ETT) and auscultation for air passing around the ETT. If air movement is not audible on auscultation (a failed CLT) there is a potential presence of laryngeal edema (LE) that may cause post-extubation airway obstruction.
  Arms: Intervention - Cuff Leak Test
Drug: Dexamethasone 4mg — Dexamethasone, will be administered to those patients who fail the CLT in the intervention arm (4mg intravenous every 6 hours for 12-24 hours). Dexamethasone belongs to a class of drugs known as corticosteroids
  Arms: Intervention - Cuff Leak Test

SUMMARY:
The COSMIC trial will be a multicentred, national, parallel-group, pragmatic vanguard pilot trial.

DETAILED DESCRIPTION:
The COSMIC trial will be a multicentred, national, parallel-group, pragmatic vanguard pilot trial in adults (≥18 years) who are mechanically ventilated in the ICU with risk factors for LE and an order to extubate has been provided by the treating physician.

The aims of this study are to assess:

1. Protocol adherence
2. Recruitment rates
3. Secondary clinical outcomes will be collected, and if feasibility criteria are met, ultimately used in the powered trial pending no major protocol adjustments (otherwise will be reported as cohort data).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 yrs. of age
* Mechanically ventilated in the ICU \
* An order to extubate has been provided by the treating physician
* Meet at least 1 criteria for risk factors for Laryngeal Edema(LE):
* Criteria 1
* Intubated for >5 days
* Criteria 2 *must fulfill category 1 and ≥1 risk factor in category 2
* Category 1

  - Intubated for >48 hours
* Category 2

  * An unplanned extubation event within the last week
  * Airway trauma secondary to an endotracheal intubation during the past week defined as one of the following:
  * More than one attempt at direct laryngoscopy
  * More than one attempt to pass the ETT
  * Charted as a traumatic intubation
* A body mass index of >30kg/m2
* An endotracheal tube greater than 8mm in a man or 7mm in a woman
* A total positive cumulative fluid balance of at least >1500ml/d x # of days admitted to ICU (eg. If admitted for 4 days, the patient will meet this criterion if they are 6L positive during their length of ICU admission)
* Physician concern about possible laryngeal edema for a reason not previously listed above. For example:
* Prone or Trendelenburg position in a recent operation
* Agitation defined as a RASS of 3+ or more or a SAS of 6 or more that may result in airway injury

Exclusion Criteria:

* Palliative care plan or plan of care does not include re-intubation, Decision to withdraw life support, or no plan for re-intubation
* Known pregnancy: Current pregnancy or up to and including 7 days postpartum
* Patients with highly suspected laryngeal injury: Burn patients, smoke inhalation injuries, blunt or penetrating trauma of the neck and airway, recent head and neck surgeries, and patients admitted with airway edema
* Known pre-existing tracheolaryngeal abnormalities: Vocal cord paralysis, tracheolaryngeal neoplasm, tracheomalasia, tracheolaryngeal stenosis, or previous head and neck surgeries
* Mechanical ventilation via a tracheostomy
* High dose steroids administered within the previous 72h (Prednisone 1mg/kg oral equivalent)
* The ICU physician believes the patient should have a CLT performed
* Patient had a failed CLT in the previous 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Protocol Adherence | 30 days
  Define a successful adherence rate as ≥75%. We will calculate the adherence as the proportion of patients that are assigned to the intervention arm following the appropriate treatment algorithm and those assigned to the control arm being extubated without a cuff leak test. As this pilot trial is ongoing, we will review adherence monthly and investigate the reasons for compliance failure. We will investigate all reasons for failure to follow the treatment algorithm in the intervention arm, failure to extubate after a patient passes a CLT in the intervention arm, or failure to extubate immediately after randomization in the control arm and report them as a protocol violation. The RC will review the RT's charting and the medication profile to determine actual compliance. RC will record all reasons for non-compliance using distinguishing clinical reasons (eg, palliation, death, consent withdrawal and errors).
Recruitment Rate | 1 Year
  Define a successful recruitment rate as enrolling three patients per centre per month over the duration of the trial. While the pilot trial is ongoing, steering committee will review recruitment weekly and the screening records monthly. If applicable, we will address barriers to enrolment to maximise recruitment. The recruitment metric will be measured and interpreted at the end of the pilot trial by calculating the mean number of recruited patients per active screening month.

SECONDARY OUTCOMES:
Proportion of patients with Clinically Significant post-extubation stridor | within 72 hours of extubation;
  Defined as the presence of an inspiratory noise following extubation that requires medical intervention such as racemic epinephrine
Proportion of patients Reintubation | within 72 hours of extubation;
  Re insertion of an endotracheal tube to maintain an airway within 72 hours for any reason (reasons for reintubation will be captured)
Proportion of patients with Post-extubation stridor | within 72 hours of extubation
  Defined as the presence of an inspiratory noise following extubation.
Proportion of patients with Emergency Surgical Airway | within 72 hours of extubation
  A procedure performed to secure the airway in patients with upper airway obstruction who could not be managed with intubation or mechanical ventilation.
ICU Mortality | Within 30 days of Randomization
  Death during Intensive Care Unit admission
Hospital Mortality | Within 30 days of Randomization
  Death during Intensive Care Unit admission
Ventilator Free Days | Within 30 Days of Randomization
  Number of days alive and free of mechanical ventilation.
ICU Length of Stay | Within 30 days of Randomization
  Number of days admitted to the ICU
Length of Stay | Within 30 days of Randomization
  Number of days admitted to hospital
Proportion of patients with Ventilator Associated Pneumonia | 30 Days from Randomization
  Pneumonia occurring more than 48 h after patients have been intubated and received mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kimberley Lewis, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (5):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States
- Canada (3):
  - Brantford General Hospital, Brantford, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Niagara Health System, Saint Catherines, Ontario
- Al-Amiri Hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandoz Canada Inc. Prescribing Information - Dexamethasone Sodium Phosphate Injection USP (4 mg/mL and 10 mg/mL Sterile Corticosteroid.
- [Background] Lewis K, Culgin S, Jaeschke R, Perri D, Marchildon C, Hassall K, Piraino T, Thabane L, Almubarak Y, Alshahrani MS, Rochwerg B, Baw B, Szczeklik W, Karachi T, Alhazzani W; GUIDE Group. Cuff Leak Test and Airway Obstruction in Mechanically Ventilated ICU Patients (COMIC): a pilot randomised controlled trial protocol. BMJ Open. 2019 Jul 19;9(7):e029394. doi: 10.1136/bmjopen-2019-029394. PMID 31326936
- [Background] Alhazzani W, Guyatt G, Alshahrani M, Deane AM, Marshall JC, Hall R, Muscedere J, English SW, Lauzier F, Thabane L, Arabi YM, Karachi T, Rochwerg B, Finfer S, Daneman N, Alshamsi F, Zytaruk N, Heel-Ansdell D, Cook D; Canadian Critical Care Trials Group. Withholding Pantoprazole for Stress Ulcer Prophylaxis in Critically Ill Patients: A Pilot Randomized Clinical Trial and Meta-Analysis. Crit Care Med. 2017 Jul;45(7):1121-1129. doi: 10.1097/CCM.0000000000002461. PMID 28459708
- [Background] Girard TD, Alhazzani W, Kress JP, Ouellette DR, Schmidt GA, Truwit JD, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Morris PE; ATS/CHEST Ad Hoc Committee on Liberation from Mechanical Ventilation in Adults. An Official American Thoracic Society/American College of Chest Physicians Clinical Practice Guideline: Liberation from Mechanical Ventilation in Critically Ill Adults. Rehabilitation Protocols, Ventilator Liberation Protocols, and Cuff Leak Tests. Am J Respir Crit Care Med. 2017 Jan 1;195(1):120-133. doi: 10.1164/rccm.201610-2075ST. PMID 27762595
- [Background] Seymour CW, Martinez A, Christie JD, Fuchs BD. The outcome of extubation failure in a community hospital intensive care unit: a cohort study. Crit Care. 2004 Oct;8(5):R322-7. doi: 10.1186/cc2913. Epub 2004 Jul 20. PMID 15469575
- [Background] Torres A, Gatell JM, Aznar E, el-Ebiary M, Puig de la Bellacasa J, Gonzalez J, Ferrer M, Rodriguez-Roisin R. Re-intubation increases the risk of nosocomial pneumonia in patients needing mechanical ventilation. Am J Respir Crit Care Med. 1995 Jul;152(1):137-41. doi: 10.1164/ajrccm.152.1.7599812.
- [Background] Frutos-Vivar F, Esteban A, Apezteguia C, Gonzalez M, Arabi Y, Restrepo MI, Gordo F, Santos C, Alhashemi JA, Perez F, Penuelas O, Anzueto A. Outcome of reintubated patients after scheduled extubation. J Crit Care. 2011 Oct;26(5):502-509. doi: 10.1016/j.jcrc.2010.12.015. Epub 2011 Mar 3. PMID 21376523
- [Background] Demling RH, Read T, Lind LJ, Flanagan HL. Incidence and morbidity of extubation failure in surgical intensive care patients. Crit Care Med. 1988 Jun;16(6):573-7. doi: 10.1097/00003246-198806000-00001. PMID 3371019
- [Background] Epstein SK, Ciubotaru RL. Independent effects of etiology of failure and time to reintubation on outcome for patients failing extubation. Am J Respir Crit Care Med. 1998 Aug;158(2):489-93. doi: 10.1164/ajrccm.158.2.9711045. PMID 9700126
- [Background] Zhou T, Zhang HP, Chen WW, Xiong ZY, Fan T, Fu JJ, Wang L, Wang G. Cuff-leak test for predicting postextubation airway complications: a systematic review. J Evid Based Med. 2011 Nov;4(4):242-54. doi: 10.1111/j.1756-5391.2011.01160.x. PMID 23672755
- [Background] Francois B, Bellissant E, Gissot V, Desachy A, Normand S, Boulain T, Brenet O, Preux PM, Vignon P; Association des Reanimateurs du Centre-Ouest (ARCO). 12-h pretreatment with methylprednisolone versus placebo for prevention of postextubation laryngeal oedema: a randomised double-blind trial. Lancet. 2007 Mar 31;369(9567):1083-9. doi: 10.1016/S0140-6736(07)60526-1. PMID 17398307
- [Background] Sutherasan Y, Theerawit P, Hongphanut T, Kiatboonsri C, Kiatboonsri S. Predicting laryngeal edema in intubated patients by portable intensive care unit ultrasound. J Crit Care. 2013 Oct;28(5):675-80. doi: 10.1016/j.jcrc.2013.05.011. Epub 2013 Jun 24. PMID 23806246
- [Background] Tadie JM, Behm E, Lecuyer L, Benhmamed R, Hans S, Brasnu D, Diehl JL, Fagon JY, Guerot E. Post-intubation laryngeal injuries and extubation failure: a fiberoptic endoscopic study. Intensive Care Med. 2010 Jun;36(6):991-8. doi: 10.1007/s00134-010-1847-z. Epub 2010 Mar 18. PMID 20237758
- [Background] Maury E, Guglielminotti J, Alzieu M, Qureshi T, Guidet B, Offenstadt G. How to identify patients with no risk for postextubation stridor? J Crit Care. 2004 Mar;19(1):23-8. doi: 10.1016/j.jcrc.2004.02.005. PMID 15101002
- [Derived] Estrada J, Armanious I, Perri D, Cook DJ, Duan EH, Bosma K, Hassall K, Marchildon C, Mehta S, Jaeschke R, Piraino T, Carayannopoulos KL, Alhazzani W, Lewis K. Cuff leak test and airway obstruction in mechanically ventilated ICU patients (COSMIC): a pilot feasibility randomized controlled trial protocol. BMJ Open. 2025 Jun 19;15(6):e096053. doi: 10.1136/bmjopen-2024-096053. PMID 40537229
- See also: Trial Website — https://www.cosmictrial.com/